CLINICAL TRIAL: NCT01279122
Title: Evaluation of Visual Outcomes of Monovision Patients Bilaterally Implanted With Nanoflex Intraocular Lenses
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovative Medical (Industry)
Responsible Party: Annie Christensen, IMEDS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARR2010-NF-IOL
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Patients Who Have Bilateral NanoFlex Implantation at Least 3 Months Previously

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nanoflex IOL (No Intervention)
  Interventions: Device: Nanoflex IOL

INTERVENTIONS:
Device: Nanoflex IOL — Patients who were implanted with the Nanoflex IOL

SUMMARY:
The purpose of this study is to look at how well you see the Nanoflex Intraocular lens placed in your eye.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age.
* Patients who have bilateral NanoFlex implantation at least 3 months previously.
* No significant ocular pathology causing DCVA to be less than 20/25 or causing significant visual loss.
* DCVA of 20/25 or better in both eyes.
* Spherical equivalent in the dominant eye to be +/-.50 or less and in the non-dominant eye to be between-1.00 and -1.87.
* Uncorrected VA in dominant eye 20/25 or better.

Exclusion Criteria:

* History of ocular trauma or prior ocular surgery (minor ocular trauma is allowed such as small superficial corneal scar not effecting vision; some prior ocular surgery is allowable so long as it has not impacted visual acuity.
* Amblyopia or strabismus, significant visual field loss, or posterior capsular opacifcation.
* Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Near Visual Acuity | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kenneth Lipstock, Richmond, Virginia, United States